CLINICAL TRIAL: NCT03089554
Title: Integration of Precision Medicine Into Cancer Therapeutics, Part 2: A Therapeutic Phase 2 Sub-study Evaluating Genomic Testing in Human Cancer and Outcomes of Targeted Therapies Recommended by an Institutional Multidisciplinary Molecular Tumor Board in Patients With Poor Prognosis Cancer
Brief Title: Evaluating Genomic Testing in Human Cancer & Outcomes of Targeted Therapies
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rachel Miller (Other)
Responsible Party: Sponsor-Investigator, Rachel Miller, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16-MULTI-19
Record Dates: First submitted 2017-03-17; First posted 2017-03-24 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Therapeutic Intervention (Experimental): Therapeutic Intervention
  Interventions: Drug: Therapeutic Intervention

INTERVENTIONS:
Drug: Therapeutic Intervention — Therapeutic Intervention

SUMMARY:
This is a substudy (Part 2) of a larger two-part clinical trial including both observational and therapeutic (interventional) cohorts to assess the progression free survival ratio of patients treated with a targeted therapy based on genomic analysis results and recommendation by the Markey Cancer Center Molecular Tumor Board (MCC MTB).

DETAILED DESCRIPTION:
This prospective, single-arm trial in patients with refractory metastatic cancer will compare the Progression Free Survival (PFS) using a treatment regimen selected by the MCC MTB with the PFS (time to tumor progression) for the most recent regimen on which the patient had experienced progression (i.e., using patients as their own control).

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically suspected or histologically confirmed solid or hematological malignancy who have undergone or will undergo genetic testing of their tumor
* Patients must have failed first-line therapy for their disease (refractory) or have no options for curative therapies.
* Patients must have either measurable or non-measurable disease.
* Age ≥18 years.
* Eastern Cooperative Oncology Group performance status ≤3.
* Patients with brain metastasis must have had treatment of their brain metastasis completed at least 1 day prior to enrollment and be on stable dose of steroids or off steroids at the time of enrollment.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with targeted therapy, in the opinion of the treating physician.
* Pregnant women are excluded from this study.
* HIV positive patients with CD4 counts below 500 OR who are not on a stable dose of antiretroviral therapy (for at least 1 month prior to registration) are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2017-04-11 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 2 years
  Proportion of patients achieving a PFS ratio ≥1.3.

CONTACTS AND LOCATIONS:
Overall Officials: RACHEL MILLER, MD, Principal Investigator — University of Kentucky
Locations (1):
- Markey Cancer Center, University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miller RW, Hutchcraft ML, Weiss HL, Wu J, Wang C, Liu J, Jayswal R, Buchanan M, Anderson A, Allison DB, El Khouli RH, Patel RA, Villano JL, Arnold SM, Kolesar JM. Molecular Tumor Board-Assisted Care in an Advanced Cancer Population: Results of a Phase II Clinical Trial. JCO Precis Oncol. 2022 Aug;6:e2100524. doi: 10.1200/PO.21.00524. PMID 36103643